CLINICAL TRIAL: NCT06243172
Title: Determining Circadian Metabolic and Behavioural Rhythms in Patients with and Without Type 2 Diabetes and Identifying the Relation to Hormone and Glucose Fluctuations, and Cognition
Brief Title: Determining Circadian Metabolic and Behavioural Rhythms in Patients with and Without Type 2 Diabetes
Acronym: Cir-D-Brain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Sponsor
Other Study IDs: H-22014311
Record Dates: First submitted 2024-01-28; First posted 2024-02-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes; Circadian Rhythm
Keywords: Type 2 Diabetes; Circadian Rhythm; Cognition; Sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Type 2 Diabetes: Individuals with type 2 diabetes
- Controls: Individuals without type 2 diabetes matched on age and body mass index

SUMMARY:
The goal of the present clinical descriptive study is to characterize and quantify the potential hormonal chronobiological differences between individuals with type 2 diabetes (T2D) and healthy age and weight-matched controls as either circadian aligned or misaligned. The investigators hypothesize that individuals with T2D have a misaligned and different circadian rhythmicity of circadian biomarkers (melatonin and cortisol) than controls, and that this difference in turn is related to 24h hormonal fluctuations, behaviour, and metabolic-, cardiac-, and cognitive parameters.

Participants will be asked to:

* fill-out a diary on eating and sleeping habits for 30 days
* wear an actigraphy and continuous glucose monitor for 10-14 days
* stay overnight at the research facility, including continuous blood sampling and polysomnography

DETAILED DESCRIPTION:
T2D is associated with cognitive dysfunction and an increased risk of developing dementia. This negative effect on cognition is worsened by T2D duration, yet the mechanisms are unknown.

Sleep disturbances increase peripheral insulin resistance, and is associated with the development of T2D, temporarily worsened cognitive function, and the development of cognitive impairment. In turn, T2D is associated with circadian misalignment (a condition where the internal physiological clock is unaligned with the external behavior). A major external signal (also known as zeitgeber) for synchronizing the internal and external clock is sleep in accordance with the day-night cycle.

Determining the circadian rhythm of an individual and whether it is aligned or misaligned is complex and can't be done by one measurement. However, melatonin and cortisol are often used as "circadian biomarkers" due to significant and well-defined circadian rhythm profiles. Another measure of the circadian phase is the timing of melatonin production under dim light conditions (dim light melatonin onset) which is an individual phase marker depending on the persons habitual time of sleep. Most studies focusing on circadian alignment in an everyday setting have used questionnaires, and to our knowledge, no studies have described 24-h circadian oscillations between individuals with T2D and healthy age and weight matched controls. Mapping these potential differences could help explain the pathophysiological mechanisms behind T2D and circadian misalignment.

The Cir-D-Brain study is a clinical descriptive study. The study comprises of an information visit, a screening visit, a midway visit (2 weeks after screening), a 24-h in-hospital day (a day between the midway visit and the final visit), and a final visit (2 weeks after the midway visit). Participants will keep a diary on eating and sleeping habits for all 30 days. At the midway visit, participants will be equipped with an actigraphy and a continuous glucose monitor. At the 24-h in-hospital day, participants will have their blood sampled every third hour for 24 hours to measure their circadian rhythm, every hour from 6 pm till 12 am to map dim light melatonin onset, and at wake-up to map cortisol awakening response. At the 24-h in-hospital day, participants will furthermore have their sleep stages measured by polysomnography. The study will include 30 participants with T2D and 30 age and BMI matched controls.

The specific objectives are:

1. To characterize and quantify the hormonal chronobiological differences between individuals with T2D and healthy matched controls measured by circadian biomarkers.
2. To relate the findings to 24-h hormonal fluctuations, different patterns in metabolism, behavioural circadian rhythms differences (sleep-wake and eating habits), sleep stages, glycaemic variability, inflammation, heart rate variability, and cognition.

ELIGIBILITY:
Inclusion Criteria:

Individuals with T2D:

* Informed and written consent.
* Clinically diagnosed diabetes mellitus type 2 for at least 5 years (diagnosed according to criteria of World Health Organization (WHO)).
* HbA1c >53 mmol/mol
* Stable medical treatment for at least 8 weeks.
* Plasma haemoglobin ≥8.00 mmol/L (male) or ≥6.4 mmol/L (female).
* Male or female participants aged 50-75 years.

Healthy matched controls:

* Informed and written consent.
* Normal haemoglobin ≥8.00 mmol/L (male) or ≥6.4 mmol/L (female).
* Male or female participants aged 50-75 years.

Exclusion Criteria:

* Body mass index (BMI) <23 kg/m2
* Receipt of any investigational medicinal product within 3 months before screening in this trial.
* Inability to perform neuropsychological tests (e.g., visual impairment or auditory impairment, or language barrier).
* Participants with mental incapacity or language barriers precluding adequate understanding or co-operation or who, in the opinion of the investigator or their general practitioner, should not participate in the trial.
* Prior or contemporary use of any kind of hypnotica within 6 months, former p.n. use of melatonin is judged by the investigator.
* Nightshift-worker.
* Known dementia or any other major disorders that in the opinion of the investigator precludes compliance with the protocol, evaluation of the results or represent an unacceptable risk for the participant's safety.
* Diagnosed sleep disorders (e.g., sleep apnoea and narcolepsy).
* Significant history of alcoholism or drug/chemical abuse as per investigator's judgement.
* Severe hypoglycaemic event during the past 6 months requiring medical assistance.
* Diagnosed diabetic retinopathy.
* Severe renal insufficiency defined as estimated glomerular filtration rate (eGFR) ≤ 30 ml/min/1.73m2 or any kind of kidney disease that in the opinion of the investigator involves an unnecessary risk for the participants.
* Cardiac problems including any of the following:

  1. Classified as being in New York Heart Association (NYHA) class III or IV.
  2. Angina pectoris (chest pain) within the last 6 months.
* Inadequately treated blood pressure at screening defined as repeated resting blood pressure outside the rage 90-150 mmHg for systolic and 50-100 mmHg for diastolic blood pressure.
* Known lung disease that in the opinion of the investigator represents an unacceptable risk for the participant's safety.
* Active or recent (≤ 12 months) malignant disease is judged by the investigator.
* For females only: Pregnancy, breast-feeding status, or intention of becoming pregnant during the trial.
* For healthy matched controls: prediabetes defined as HbA1c between 42-47 mmol/mol

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, Steno Diabetes Center Copenhagen out-patient clinic, community sample
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Melatonin oscillations (amplitude, peak, mesor, phase, period length (TAU)) | 24-hour in-hospital day, blood samples taken every third hour for 24 hours (9 timepoints in total)
  Blood samples
Cortisol oscillations (amplitude, peak, mesor, phase, period length (TAU)) | 24-hour in-hospital day, blood samples taken every third hour for 24 hours (9 timepoints in total)
  Blood samples

SECONDARY OUTCOMES:
Dim light melatonin onset | 24-hour in-hospital day, blood samples taken every hour from 18:00 until 00:00 (7 timepoints in total)
  Blood samples (pg/ml)
Phase angle (time between dim light melatonin onset and sleep) | 24-hour in-hospital day, blood samples taken every hour from 18:00 until 00:00 (7 timepoints in total)
  Blood samples
Cortisol awakening response | 24-hour in-hospital day, blood samples taken at wake up, and 15-, 30-, and 60-minutes post-wake up
  Blood samples (pg/ml)
Diary on sleeping habits | 30 days
  Expanded Consensus Sleep Diary (time in bed, time to fall asleep, number of awakenings and durations, time of final awakening, time to get out of bed, total sleep time, sleep quality, daytime sleepiness, number of naps and duration, number and last time of alcohol consumption, number and last time of coffein consumption, use of sleep medicine)
Diary on eating window | 30 days
  The eating window (initiation of first consumption and termination of last consumption of food)
Glycaemic variability | 10-14 days
  Continuous glucose monitor (amplitude (mmol/L), frequency, and duration of the fluctuation, mean glucose (mmol/L), time in range, time in hyperglycemic and hypoglycemic range, area under the curve)
Sleep and waking states | 10-14 days
  Actrigraph worn on the wrist of the non-dominant hand (acceleration at different times)
Heart rate variability (fluctuations in time intervals between adjacent heart beats) | 24-hour in-hospital day
  Measured continuously by the polysomnograph (ms)
Sleep architecture | 24-hour in-hospital day
  Polysomnography (minutes and percentages). Sleep stages (N1, N2, N3, rapid eye movement (REM)), total time asleep, sleep latency, REM sleep latency, arousals, awakenings, total sleep efficiency.
Cognition (verbal memory) | 24-hour in-hospital day
  Rey Auditory Verbal Learning Test (RAVLT)
Cognition (psychomotor speed and executive function) | 24-hour in-hospital day
  Trail Making Test (TMT) part A and B ), Symbol Digit Modalities Test (SDMT)
Cognition (executive function) | 24-hour in-hospital day
  WAIS-III Letter-Number Sequencing test, Verbal fluency test (letters S and D)
Cognition (sustained attention) | 24-hour in-hospital day
  Rapid Visual Processing (RVP) test from the Cambridge Neuropsychological Test Automated Battery (CANTAB)
Cognition (verbal IQ) | 24-hour in-hospital day
  Danish Adult Reading Test (DART) (equivalent to the National Adult Reading Test; NART)
Insulin oscillations (amplitude, peak, mesor, phase, period length (TAU)) | 24-hour in-hospital day, blood samples taken every third hour for 24 hours (9 timepoints in total)
  Blood samples.
C-peptide oscillations (amplitude, peak, mesor, phase, period length (TAU)) | 24-hour in-hospital day, blood samples taken every third hour for 24 hours (9 timepoints in total)
  Blood samples.
TSH oscillations (amplitude, peak, mesor, phase, period length (TAU)) | 24-hour in-hospital day, blood samples taken every third hour for 24 hours (9 timepoints in total)
  Blood samples.
Glucose oscillations (amplitude, peak, mesor, phase, period length (TAU)) | 24-hour in-hospital day, blood samples taken every third hour for 24 hours (9 timepoints in total)
  Blood samples.
Glucagon oscillations (amplitude, peak, mesor, phase, period length (TAU)) | 24-hour in-hospital day, blood samples taken every third hour for 24 hours (9 timepoints in total)
  Blood samples.
Glucagon-like peptide-1 (GLP-1) oscillations (amplitude, peak, mesor, phase, period length (TAU)) | 24-hour in-hospital day, blood samples taken every third hour for 24 hours (9 timepoints in total)
  Blood samples.

OTHER OUTCOMES:
Chronotype (diurnal preference) | At screening
  Morningness-Eveningness Questionnaire (scoring)
Sleep apnea | 24-hour in-hospital day
  Apnea-hypopnea index (events/hour)
Blood pressure variations | 24-hour in-hospital day
  Measured continuously by the polysomnograph (mmHg)
Cardiovascular autonomic neuropathy | At screening
  Assessed from three standard cardiovascular autonomic reflex tests: lying-to-standing test, deep breathing test, and Valsalva manoeuvre

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Rungby, MD, DMSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No